CLINICAL TRIAL: NCT03048071
Title: Morbimortality of Contegra Duct Replacements Versus Homografts in Pulmonary Position: a Comparative Study
Brief Title: Morbimortality of Contegra Duct Replacements Versus Homografts in Pulmonary Position
Status: Completed | Type: Observational
Sponsor: Pierre Wauthy (Other)
Responsible Party: Sponsor-Investigator, Pierre Wauthy, Head of clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-Conegra vs homografts
Record Dates: First submitted 2017-02-02; First posted 2017-02-09 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Congenital Heart Disease
Keywords: Contegra; Homograft
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Homograft in pulmonary position replacement: All patients having had the replacement of an homograft in pulmonary position between January 1999 and October 2016, within the Queen Fabiola Children Hospital of Brussels, Belgium.
  Interventions: Other: Data collection within medical files
- Contegra conduct replacement: All patients having had the replacement of a Contegra conduct between January 1999 and October 2016, within the Queen Fabiola Children Hospital of Brussels, Belgium.
  Interventions: Other: Data collection within medical files

INTERVENTIONS:
Other: Data collection within medical files — Data collection within medical files

SUMMARY:
Congenital heart diseases are nowadays frequently treated in newborns. These congenital heart defects can directly affect the right ventricular ejection tract (RVOT), or sometimes indirectly, when the left ventricular ejection tract (LVOT) is replaced by the ROVT in a Ross operation. Originally introduced by Ross and Somerville in 1966, the reconstruction of ROVT by valved homografts is since then widely used.Pulmonary and aortic homografts then constituted the gold standard in conduit replacement between the right ventricle and the pulmonary artery (VD-AP).

The increasing demand for homografts currently induces a shortage and unmet demands. This lack of availability, and the durability of homografts in young patients, has encouraged the search for alternative conducts.For example, in 1999, Medtronic® put a bovine jugular vein xenograft (VJB) on the market, the Contegra® conduct, as alternative for the homograft for RVOT reconstruction. This duct naturally has a central valve with three valvules, and there is on both sides of the valve a generous duct length allowing unique adaptation options. This conduit, however, is not perfect.

Whether using Contegra® ducts or homografts, replacement is inevitable. The aim of this study is to compare operative morbidity and mortality when replacing Contegra® or homograft.

DETAILED DESCRIPTION:
Congenital heart diseases are nowadays frequently treated in newborns. These congenital heart defects can directly affect the right ventricular ejection tract (RVOT), or sometimes indirectly, when the left ventricular ejection tract (LVOT) is replaced by the ROVT in a Ross operation. Originally introduced by Ross and Somerville in 1966, the reconstruction of ROVT by valved homografts is since then widely used. The technique became particularly popular from the mid-1980s, through the routine use of cryopreservation. Pulmonary and aortic homografts then constituted the gold standard in conduit replacement between the right ventricle and the pulmonary artery (VD-AP). Early failure of homografts is mainly due to early calcifications. Lung homografts are, however, less prone to obstructions and calcifications than aortic homografts but are not readily available, particularly in small sizes (10-18mm).

The increasing demand for homografts currently induces a shortage and unmet demands. This lack of availability, and the durability of homografts in young patients, has encouraged the search for alternative conducts. For example, in 1999, Medtronic® put a bovine jugular vein xenograft (VJB) on the market, the Contegra® conduct, as alternative for the homograft for RVOT reconstruction. This duct naturally has a central valve with three valvules, and there is on both sides of the valve a generous duct length allowing unique adaptation options. It is stored in a glutaraldehyde solution in concentrations sufficient enough to make it non-antigenic, yet low enough to maintain the flexibility of the tissue.This conduit has many advantages: 1) Immediate availability 2) Available size range from 12 to 22mm internal diameter 3) Possibility of adaptation to morphology and easily suturable 4) Good hemodynamics 5) No need for proximal or distal extension 6) lower cost than homograft and 7) non-antigenicity.

This conduit, however, is not perfect. On the one hand, it has no growth potential and therefore risks becoming too small and no longer suitable as the child develops. This problem is particularly encountered in small patients, in whom ducts less than 16mm in diameter have been implanted, and is not specific to the duct in VJB. On the other hand, there is a source of failure specific to the Contegra® prosthesis. These are the stenoses at the level of the distal anastomosis between the duct and the pulmonary artery. Several mechanisms explain this distal stenosis: 1) hypoplasia or distal stenosis of the branches of the pulmonary artery, 2) difference in size between the duct and the pulmonary artery being too important, 3) the surgical technique , 4) immunological and inflammatory reactions, 5) neointimal proliferation, 6) thrombi formation. The most likely cause is multifactorial, with a combination of factors cited above.

Prior et al proposed an operative protocol for reducing the distal stenosis rate. With this protocol distal stenosis has become a rare complication but there are still situations in which the VJB conduit needs to be replaced.

Therefore, whether using Contegra® ducts or homografts, replacement is inevitable. The aim of this study is to compare operative morbidity and mortality when replacing Contegra® or homograft.

ELIGIBILITY:
Inclusion Criteria:

* All patients having had the replacement of a Contegra conduct, or the replacement of an homograft in pulmonary position, between January 1999 and October 2016, within the Queen Fabiola Children Hospital of Brussels, Belgium.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients having had the replacement of a Contegra conduct, or the replacement of an homograft in pulmonary position, between January 1999 and October 2016, within the Queen Fabiola Children Hospital of Brussels, Belgium.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Age | 18 years
  Age of the child when replacement surgery is performed
Length of time between placement surgery and replacement surgery | 18 years
  Length of time between the placement of the homograft/Contegra and its replacement
Weight | 18 years
  Weight of the child before replacement surgery
Sex | 18 years
  Sex of the child
Homograft/contegra position (anatomic/extra anatomic) | 18 years
  Anatomic or extra anatomic position
Co-intervention (yes/no) | 18 years
  Presence of another surgical intervention during the homograft/contegra replacement surgery
Total duration of intervention | 18 years
  Total duration of the replacement surgery
Total duration of extra corporeal circulation | 18 years
  Total duration of extra corporeal circulation during the replacement surgery
Aortic clampage duration | 18 years
  Total duration of aortic clampage duration during the replacement surgery
Duration of circulatory arrest | 18 years
  Total duration of circulatory arrest during the replacement surgery
Presence of perioperatory complications (yes/no) | 18 years
  Presence of perioperatory complications (yes/no) during the replacement surgery
PRISM Score | 18 years
  Pediatric Risk of Mortality score, ad defined by the pediatric ICU in post-replacement surgery care
Inotropic duration | 18 years
  Inotropic duration in post-replacement surgery care
Extubation day | 18 years
  Number of days between the surgery and the extubation in post-replacement surgery care
Length of stay in ICU | 18 years
  Number of days in ICU after replacement surgery
Length of hospitalisation after replacement surgery | 18 years
  Length of hospitalisation after replacement surgery
Cause of death | 18 years
  Cause of death after replacement surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Poinot, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ross DN. Replacement of aortic and mitral valves with a pulmonary autograft. Lancet. 1967 Nov 4;2(7523):956-8. doi: 10.1016/s0140-6736(67)90794-5. No abstract available. PMID 4167516
- [Background] Ross DN, Somerville J. Correction of pulmonary atresia with a homograft aortic valve. Lancet. 1966 Dec 31;2(7479):1446-7. doi: 10.1016/s0140-6736(66)90600-3. No abstract available. PMID 4163445
- [Background] Boethig D, Goerler H, Westhoff-Bleck M, Ono M, Daiber A, Haverich A, Breymann T. Evaluation of 188 consecutive homografts implanted in pulmonary position after 20 years. Eur J Cardiothorac Surg. 2007 Jul;32(1):133-42. doi: 10.1016/j.ejcts.2007.02.025. Epub 2007 Apr 18. PMID 17446081
- [Background] Brown JW, Ruzmetov M, Rodefeld MD, Vijay P, Darragh RK. Valved bovine jugular vein conduits for right ventricular outflow tract reconstruction in children: an attractive alternative to pulmonary homograft. Ann Thorac Surg. 2006 Sep;82(3):909-16. doi: 10.1016/j.athoracsur.2006.03.008. PMID 16928507
- [Background] Hickey EJ, McCrindle BW, Blackstone EH, Yeh T Jr, Pigula F, Clarke D, Tchervenkov CI, Hawkins J; CHSS Pulmonary Conduit Working Group. Jugular venous valved conduit (Contegra) matches allograft performance in infant truncus arteriosus repair. Eur J Cardiothorac Surg. 2008 May;33(5):890-8. doi: 10.1016/j.ejcts.2007.12.052. Epub 2008 Mar 4. PMID 18313324
- [Background] Corno AF, Hurni M, Griffin H, Galal OM, Payot M, Sekarski N, Tozzi P, von Segesser LK. Bovine jugular vein as right ventricle-to-pulmonary artery valved conduit. J Heart Valve Dis. 2002 Mar;11(2):242-7; discussion 248. PMID 12000167
- [Background] Fiore AC, Brown JW, Turrentine MW, Ruzmetov M, Huynh D, Hanley S, Rodefeld MD. A bovine jugular vein conduit: a ten-year bi-institutional experience. Ann Thorac Surg. 2011 Jul;92(1):183-90; discussion 190-2. doi: 10.1016/j.athoracsur.2011.02.073. Epub 2011 May 6. PMID 21549348
- [Background] Urso S, Rega F, Meuris B, Gewillig M, Eyskens B, Daenen W, Heying R, Meyns B. The Contegra conduit in the right ventricular outflow tract is an independent risk factor for graft replacement. Eur J Cardiothorac Surg. 2011 Sep;40(3):603-9. doi: 10.1016/j.ejcts.2010.11.081. Epub 2011 Feb 19. PMID 21339072
- [Background] Yong MS, Yim D, d'Udekem Y, Brizard CP, Robertson T, Galati JC, Konstantinov IE. Medium-term outcomes of bovine jugular vein graft and homograft conduits in children. ANZ J Surg. 2015 May;85(5):381-5. doi: 10.1111/ans.13018. Epub 2015 Feb 23. PMID 25708132
- [Background] Prior N, Alphonso N, Arnold P, Peart I, Thorburn K, Venugopal P, Corno AF. Bovine jugular vein valved conduit: up to 10 years follow-up. J Thorac Cardiovasc Surg. 2011 Apr;141(4):983-7. doi: 10.1016/j.jtcvs.2010.08.037. Epub 2010 Sep 29. PMID 20884023
- [Background] Shebani SO, McGuirk S, Baghai M, Stickley J, De Giovanni JV, Bu'lock FA, Barron DJ, Brawn WJ. Right ventricular outflow tract reconstruction using Contegra valved conduit: natural history and conduit performance under pressure. Eur J Cardiothorac Surg. 2006 Mar;29(3):397-405. doi: 10.1016/j.ejcts.2005.11.040. Epub 2006 Jan 24. PMID 16439155
- [Background] Holmes AA, Co S, Human DG, Leblanc JG, Campbell AI. The Contegra conduit: Late outcomes in right ventricular outflow tract reconstruction. Ann Pediatr Cardiol. 2012 Jan;5(1):27-33. doi: 10.4103/0974-2069.93706. PMID 22529597
- [Background] Corno AF, Mickaily-Huber ES. Comparative computational fluid dynamic study of two distal Contegra conduit anastomoses. Interact Cardiovasc Thorac Surg. 2008 Feb;7(1):1-5. doi: 10.1510/icvts.2007.162412. Epub 2007 Sep 28. PMID 17905782
- [Derived] Poinot N, Fils JF, Demanet H, Dessy H, Biarent D, Wauthy P. Pulmonary valve replacement after right ventricular outflow tract reconstruction with homograft vs Contegra(R): a case control comparison of mortality and morbidity. J Cardiothorac Surg. 2018 Jan 17;13(1):8. doi: 10.1186/s13019-018-0698-5. PMID 29343297